CLINICAL TRIAL: NCT06992063
Title: Evaluation of Post-dural Puncture Headache in Female Patients Undergoing Obstetric and Non-obstetric Surgery
Status: Recruiting | Type: Observational
Sponsor: Duzce University (Other)
Responsible Party: Principal Investigator, Özlem Ersoy Karka, Assistant Professor, Duzce University
Other Study IDs: drozlemersoy7
Record Dates: First submitted 2025-04-21; First posted 2025-05-28 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Post-Dural Puncture Headache
MeSH Terms: conditions — Post-Dural Puncture Headache | interventions — Anesthesia, Spinal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Obstetric: 56 female obstetric patients undergoing spinal anesthesia
  Interventions: Procedure: Spinal anesthesia
- Non-obstetric: 56 female non-obstetric patients undergoing spinal anesthesia
  Interventions: Procedure: Spinal anesthesia

INTERVENTIONS:
Procedure: Spinal anesthesia — In both groups patients will undergo spinal anesthesia and be followed intra- and postoperatively in the context of postdural puncture headache

SUMMARY:
The goal of this observational study is to compare the incidence, severity, and potential risk factors for Post-dural Puncture headaches (PDPH) in obstetric and non-obstetric female patients undergoing spinal anesthesia. The main questions it aims to answer are:

Are there differences between these two groups? Are there contributing factors? Researchers will compare obstetric and non-obstetric patients to see if pregnancy affects female patients in context of PDPH.

Participants will be monitored periodically for PDPH development. The frequency and severity of headaches will be assessed using the Numerical Rating Scale (NRS) and Wong-Baker Scale. Additionally, the need for medical consultations and any complications arising from PDPH will be recorded.

DETAILED DESCRIPTION:
After obtaining informed consent, eligible patients will be included in the study. Demographic data and headache history will be recorded, and preoperative anxiety levels will be assessed using the State-Trait Anxiety Inventory (STAI).

In the operating room, patients will be monitored with electrocardiography, pulse oximetry, non-invasive blood pressure, and Pleth Variability Index (PVI) sensors. Baseline measurements, including peak heart rate (HR), peripheral oxygen saturation (SpO2), systolic (SBP) and diastolic blood pressure (DBP), mean arterial pressure (MAP) and PVI will be recorded. Measurements will be repeated at five-minute intervals for the first 30 minutes of the operation and at 15-minute intervals thereafter.

Following spinal anesthesia, procedural details such as the experience level of the practitioner, patient positioning, needle brand, type and size, number of attempts, puncture level, and anesthetic dose will be documented.

Patients will be monitored periodically for PDPH development. The frequency and severity of headaches will be assessed using the Numerical Rating Scale (NRS) and Wong-Baker Scale. Additionally, the need for medical consultations and any complications arising from PDPH will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18-65 years undergoing surgery under spinal anesthesia
* Patients classified as ASA I or II according to the American Society of Anesthesiologists (ASA) classification

Exclusion Criteria:

* ASA III and above patients
* Patients requiring Intensive Care Unit (ICU) admission
* Patients with mental retardation
* Patients with communication difficulties (e.g., hearing loss, speech impediments, language barriers)
* Conversion to general anesthesia due to pain after spinal anesthesia
* Emergency surgeries

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Obstetric and non-obstetric female patients undergoing spinal anesthesia
Sampling Method: Probability Sample
Enrollment: 112 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Headache development for patients who can read and write | 1 time preoperatively in the premedication unit, 1 time per hospitalization day postoperatively up to 7 days and on the 7th, 14th, 21st, and 30th postoperative days after discharge by phone call
  Development of post-dural puncture headache will be assessed using the Numerical Rating Scale (NRS) NRS is a scale between 0 (no pain) and 10 (most severe pain the patient has ever felt in is/her life). It is suitable for patients who can read and write.
Headache development for patients who cannot read and write | 1 time preoperatively in the premedication unit, 1 time per hospitalization day postoperatively up to 7 days and on the 7th, 14th, 21st, and 30th postoperative days after discharge by phone call
  Development of post-dural puncture headache will be assessed using Wong-Baker Faces Pain Rating Scale.
  The Wong-Baker Faces Pain Rating Scale is a tool that uses a combination of faces and words to help a person effectively communicate the severity of their physical pain. It is suitable for patients who cannot read and write.

SECONDARY OUTCOMES:
Preoperative anxiety | 1 time preoperatively in the premedication room
  Preoperative anxiety levels will be assessed using the State-Trait Anxiety Inventory (STAI).
  STAI is a test to assess both state and trait anxiety separately. Each type of anxiety has its own scale of 20 different questions that are scored.
  Scores range from 20 to 80, with higher scores correlating with greater anxiety.
Contributing factors: The experience level of the practitioner | 1 time intraoperatively
  The experience level of the practitioner will be recorded once when dural puncture is performed.
  It will be assessed as "1-3 years, 3-5 years, 5-10 years and over 10 years of practice".
Contributing factors: The patient positioning | 1 time intraoperatively
  The patient position will be recorded once when dural puncture is performed. It will be assessed as "sitting position, lateral decubitus or prone position".
Contributing factors: The needle factors | 1 time intraoperatively
  Needle brand, type and size will be recorded once when dural puncture is performed.
Contributing factors: The number of puncture attempts | 1 time intraoperatively
  The number of attempts will be recorded once when dural puncture is performed.
Contributing factors: The puncture level | 1 time intraoperatively
  The vertebral level of dural puncture will be recorded once when dural puncture is performed.
Contributing factors: The anesthetic dose | 1 time intraoperatively
  The total dose of local anesthetic drug will be recorded once when spinal anesthesia is performed.

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Ersoy Karka, Study Chair — Düzce University Faculty of Medicine
Locations (1):
- Duzce University Faculty of Medicine, Düzce, Düzce, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided